CLINICAL TRIAL: NCT03078881
Title: LUSTRO: A Clinical Assessment Study in Crigler-Najjar Syndrome
Brief Title: Clinical Assessment Study in Crigler-Najjar Syndrome
Acronym: LUSTRO
Status: Completed | Type: Observational
Sponsor: Audentes Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: AT342-01
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Crigler-Najjar Syndrome
MeSH Terms: conditions — Crigler-Najjar Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a Pre-Phase 1 prospective, non-interventional clinical assessment study to evaluate Crigler-Najjar syndrome subjects requiring daily phototherapy, aged 1 year and older.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has a diagnosis of Crigler-Najjar syndrome resulting from a confirmed mutation in the UGT1A1 gene
* Subject is aged equal or greater than 1 year of age
* Subject receives daily phototherapy for a minimum of 6 hours within a 24-hour period (daily illumination time)

Exclusion Criteria:

* Subject is currently participating in an interventional study or has received gene or cell therapy
* Subject has received a whole liver, partial liver, or hepatocyte transplant; or subject has a liver transplant scheduled within the planned participation period of this study
* Subject has significant cholestatic disease, in the opinion of the investigator
* Subject is receiving phenobarbital or other known inducer of UGT1A1 within 30 days of screening
* Subject has any clinically significant underlying liver disease (other than Crigler-Najjar syndrome), in the opinion of the investigator
* Subject has a history of, or currently has, a clinically important condition other than Crigler-Najjar syndrome, in the opinion of the investigator

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll Crigler-Najjar syndrome subjects aged equal or greater than 1 year of age requiring daily phototherapy.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Characterize the disease course and natural history of subjects with Crigler-Najjar syndrome | Up to 2 years
Assess variation in bilirubin levels over the course of the study and the variation of bilirubin levels over a 24-hr period | Up to 2 years
Assess phototherapy usage over the course of the study | Up to 2 years

SECONDARY OUTCOMES:
Assess the humanistic and clinical burden of disease in Crigler-Najjar subjects and caregivers as measured by PedsQL | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Suyash Prasad, MBBS, MRCP,MRCPCH, FFPM, Study Director — Audentes Therapeutics
Locations (4):
- United States (2):
  - Children's Hospital at Montefiore, The Bronx, New York
  - Clinic for Special Children, Strasburg, Pennsylvania
- Shaare Zedek Medical Center, Jerusalem, Israel
- King's College Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No